CLINICAL TRIAL: NCT01306357
Title: Evaluation De L'Observance Globale Et De La Duree De Traitement Par Zomacton® Avec Le Stylo Transjecteur Zomajet® Etude Pharmaco-Epidemiologique Observationnelle Longitudinale Prospective
Brief Title: Evaluation of Overall Compliance and Duration of Zomacton® Treatment With the Zomajet® Needle-free Device
Acronym: ZOMAJET
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: RZO 01
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2012-02

CONDITIONS: Turner's Syndrome; Human Growth Hormone Deficiency
Keywords: Turner's syndrome; somatropin; human growth hormone deficiency
MeSH Terms: conditions — Turner Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Zomacton® with Zomajet® needle-free device: Zomacton® 4 mg delivered by percutaneous transjection (needle-free) using the Zomajet® 2 Vision device or Zomacton® 10 mg delivered by percutaneous transjection (needle-free) using the Zomajet® Vision X needle-free device.
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — 4 mg or 10 mg delivered by needle-free device
  Other Names: human growth hormone; Zomacton

SUMMARY:
The purpose of this strictly observational, prospective, longitudinal study is to evaluate with sufficient precision the rate of overall treatment compliance from one year to 3 years of follow-up of the patients.

Somatotropin is indicated in the long-term treatment of children with growth retardation related to a deficiency in secretion of growth hormone and in the long-term treatment of growth retardation related to Turner's syndrome confirmed by chromosomal analysis. These are the two indications of Zomacton® 4 mg and 10 mg injection solution.

The use of the Zomajet® needle-free device (Zomajet® 2 Vision, reserved for the administration of Zomacton® 4 mg or of the Zomajet® Vision X needle-free device, reserved for the administration of Zomacton® 10 mg), allows the product to be administered by percutaneous transjection (needle-free) and can be used by the child directly or by the family after an initial training.

In April 2004, the CEPP (Commission for the Evaluation of Products and Services) requested a follow-up of the cohort of patients using the Zomajet® 2 Vision system measuring the compliance and duration of use of the device.

The number of patients initiated on Zomacton treatment using the Zomajet® needle-free device is estimated to 30. Over a period of inclusion of 3 years, we therefore estimate that 90 patients will be treated. In the cohort studied the patients will be followed-up for 1 year at least and for 3 years at the maximum.

The rate of treatment compliance will be evaluated according to the ratio of the actual duration of administration over the total duration recommended by the physician during the observation period.

ELIGIBILITY:
Inclusion Criteria:

* Growth hormone deficiency
* Turner's syndrome

Exclusion Criteria:

* Patients who do not meet the criteria in the treatment Information Sheet

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients who meet the criteria of the Treatment Information Sheet (growth hormone deficiency or Turner's syndrome) for which treatment is initiated with Zomacton® 4 mg using the Zomajet® 2 Vision needle-free device or with Zomacton® 10 mg using the Zomajet® Vision X.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2007-09; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Overall treatment compliance | up to three years

SECONDARY OUTCOMES:
Description of the auxological and biochemical characteristics of the population at inclusion (notably the exploration of GH deficiency, the height, the difference in height from the average in SD, the rate of growth prior to treatment) | Baseline (day 0)
Description of the Dosages of Growth Hormone and way of use of needle-free device | up to 3 years
Description of the evolution of the auxological and biochemical parameters (gain in height in SD, growth rate, IGF-1 if available) | Baseline (Day 0), up to three years
Average Duration of Treatment | up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (17):
- France (17):
  - Investigational site, Angers
  - Investigational site, Bordeaux
  - Investigational site, Brive-la-Gaillarde
  - Investigational site, Hyères
  - Investigational site, Juan-les-Pins
  - Investigational site, Le Mans
  - Investigational site, Lille
  - Investigational site, Lisieux
  - Investigational site, Montivilliers
  - Investigational site, Montpellier
  - Investigational site, Nice
  - Investigational site, Nieul-sur-Mer
  - Investigational site, Paris
  - Investigational site, Puyricard
  - Investigational site, Tarbes
  - Investigational site, Toulon
  - Investigational site, Toulouse